CLINICAL TRIAL: NCT01535131
Title: Furlow Palatoplasty With Tensor Tenopexy for Otitis Media
Brief Title: Furlow Palatoplasty With Tensor Tenopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Cuneyt M. Alper, Professor of Otolaryngology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO11060248; R01DC011524 (NIH)
Record Dates: First submitted 2012-02-07; First posted 2012-02-17 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Otitis Media; Cleft Palate
Keywords: otitis media; cleft palate
MeSH Terms: conditions — Otitis Media; Cleft Palate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Furlow palatoplasty (Active Comparator): standard procedure
  Interventions: Procedure: palatoplasty
- modified Furlow palatoplasty (Experimental): standard procedure plus modification
  Interventions: Procedure: palatoplasty

INTERVENTIONS:
Procedure: palatoplasty — procedure to close cleft palate

SUMMARY:
This study compares a standard method for palate repair (the Furlow palatoplasty) with a modification of that method to determine which, if either, is more effective in reducing the duration of middle-ear disease (fluid in the ear) in cleft palate patients.

DETAILED DESCRIPTION:
Almost all infants and young children who were born with a cleft palate (with or without a cleft lip) have middle-ear disease and this condition can last into late childhood and early adolescence. The type of middle-ear disease that usually occurs in cleft palate patients is not associated with pain or symptoms, but the fluid in the middle-ear causes poor hearing and sometimes problems with balance.

Past studies show that the middle-ear disease in infants and children with cleft palate is caused by their inability to open a natural tube that connects the back of the nose with the middle-ear (called the Eustachian tube). Opening the Eustachian tube is required to keep the pressure in the middle-ear equal to that of the atmosphere which prevents fluid from building up in the middle-ear. For this reason, middle-ear disease is usually treated by placing a small plastic tube in the eardrum which keeps the middle-ear pressure and pressure in the room (atmospheric pressure) equal even when the Eustachian tube fails to open. However, the disease often returns when the plastic tube becomes blocked or falls out and a new tube needs to be placed in the eardrum. The actions of two small muscles, the levator veli palatini (LVP) muscle and the tensor veli palatini (TVP) muscle combine to open the Eustachian tube and the LVP muscle plays a role in raising the palate during speech, swallowing and other activities. Both muscles run through the soft palate. In children with cleft palate, the usual position, orientation and function of both of these muscles are abnormal and few surgical procedures for palate repair focus on re-establishing a more "normal" orientation and attachment of these muscles.

One well accepted method for repair of the palate, the Furlow palatoplasty is the standard procedure used by the two cleft palate surgeons involved in this study. During the Furlow palatoplasty the attachment of the TVP muscle is cut. Recently, a modification of the Furlow palatoplasty, called a tensor tenopexy, has been described that involves attaching the cut part of the TVP muscle to a bony hook in the soft palate in an effort to improve Eustachian tube function and lead to less middle-ear disease. One small study presented results suggesting that middle-ear disease was cured at an earlier age in those cleft palate patients who had their palates repaired using the modified Furlow procedure when compared to a number of other methods of palate repair, but these comparisons did not include the standard Furlow procedure. However, the design of that study was poor and the possible benefits of this small modification in the surgical procedure with respect to middle-ear disease need to be evaluated in a more formal study. Because the surgical procedures for the Furlow palatoplasty and the modified Furlow procedure are identical with the exception of the addition of anchoring the cut muscle attachment, a study of these two procedures will allow us to determine if the modified procedure does or does not improve middle-ear disease at an earlier age in patients with cleft palate.

ELIGIBILITY:
Inclusion Criteria:

* cleft palate with or without cleft lip classified as Veau I through IV
* parental consent for procedure
* patients assigned to Drs. Losee, Davit, Grundwaldt, or Goldstein for palatoplasty
* children up to 15 months of age who have not had palatoplasty but have tympanostomy tubes

Exclusion Criteria:

* patients with syndromic clefts or genetic abnormalities

Max Age: 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2012-02-28 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
hearing status | 3-year visit
  results of audiometric testing
otitis media status | 3 years of age
  diagnosis of OM, presence/absence of ventilation tubes at time of 3-year visit
Eustachian tube function (ETF) measures | 3-year visit
  ETF test results

SECONDARY OUTCOMES:
Pittsburgh Weighted Speech Score | 3 years of age
  obtained as standard of care
nasalence ratio | 3 years of age
  obtained as standard of care
McKay-Kummer SMAP test | 3 years of age
  obtained as standard of care
duration of speech therapy | by age 7 years
need for revision palatoplasties | by 7 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Cuneyt M Alper, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No